CLINICAL TRIAL: NCT07028008
Title: Clinical Study to Evaluate the Safety and Efficacy of Autologous Tumor-infiltrating Lymphocyte (CT-SP) in Patients With Refractory Melanoma Who Failed to Immune Checkpoint Inhibitors
Brief Title: Evaluate the Safety and Efficacy of Autologous Tumor-infiltrating Lymphocyte in Patients With Refractory Melanoma Who Failed to Immune Checkpoint Inhibitors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-06-022
Record Dates: First submitted 2025-06-10; First posted 2025-06-19 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Melanoma
Keywords: melanoma; TIL
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tumor-infiltrating lymphocyte (TIL) therapy (Experimental): 1~100 x 10 9 cells, 1time, IV
  Interventions: Biological: tumor-infiltrating lymphocyte (TIL)

INTERVENTIONS:
Biological: tumor-infiltrating lymphocyte (TIL) — tumor-infiltrating lymphocyte (TIL): CT-SP 1~100 x10 9 cells

SUMMARY:
For cancer patients who have failed conventional chemotherapy or are inoperable, targeted therapies-which block specific proteins involved in tumor growth-and immunotherapies-which activate T cells around the tumor to induce tumor cell death-have emerged as powerful treatment options. These therapies often result in longer survival with fewer side effects compared to traditional chemotherapy. However, a significant proportion of patients do not respond to either targeted therapies or immunotherapies, and treatment options for these individuals remain extremely limited.

One of the most notable immunotherapies, immune checkpoint inhibitors, works by blocking immune checkpoint proteins (such as PD-1 and CTLA-4) to activate T cells within the tumor microenvironment, thereby enabling them to attack cancer cells. This approach has demonstrated remarkable efficacy in various solid tumors, including melanoma. Nonetheless, for many patients with immunologically "cold" tumors characterized by low infiltration of T cells, these therapies show low objective response rates, indicating the need for more proactive treatment strategies.

In this study, we aim to administer the tumor-infiltrating lymphocyte (TIL) therapy CT-SP to patients with refractory melanoma, primarily to assess safety, and further to evaluate its anti-tumor efficacy by examining improvements in objective response rate (ORR) and progression-free survival (PFS). If this advanced regenerative clinical study demonstrates that CT-SP is both safe and effective, it could offer a powerful new treatment option for patients with refractory melanoma in Korea.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥19 and ≤80 years at the time of informed consent.
2. Histologically or cytologically confirmed melanoma, classified as refractory/unresponsive Stage IIIc or IV after failure of prior immune checkpoint inhibitor therapy.
3. At least one measurable and evaluable lesion as defined by RECIST version 1.1.
4. ECOG performance status of 0 or 1.
5. Estimated life expectancy ≥12 weeks.
6. Ability to undergo tumor tissue biopsy for the purpose of producing a sufficient quantity of autologous tumor-infiltrating lymphocytes (CT-SP).

   * Willingness to undergo tissue collection procedures after enrollment in the study.
   * For surgical specimens: at least one lesion with a minimum diameter of 1 cm. For biopsy samples: a minimum of 20-25 tissue fragments must be obtainable.
7. Adequate organ function as defined by the following laboratory values (up to two retests permitted; transfusions or medical correction allowed):

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute Neutrophil Count (ANC) ≥ 1,500/μL
   * Absolute Lymphocyte Count (ALC) ≥ 500/μL
   * Platelet count ≥ 100,000/μL
   * Serum creatinine clearance (estimated by Cockcroft-Gault) ≥ 50 mL/min
   * Total bilirubin ≤ 2.0 mg/dL
   * AST and/or ALT ≤ 3 × ULN (≤ 5 × ULN if liver metastasis is present)
8. Subjects of childbearing potential must agree to use acceptable contraceptive methods during the study, including but not limited to:

   Complete abstinence, Sterilization (patient or partner), Intrauterine device, Hormonal contraception, Barrier methods (e.g., condom + spermicide, diaphragm)
9. Written informed consent voluntarily provided before any study-specific procedures are conducted.

Exclusion Criteria:

1. History of solid organ transplantation.
2. Diagnosis of another malignancy within the past 5 years, except for adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or non-invasive cervical cancer.
3. History of active or latent tuberculosis infection within 1 year prior to screening (except for those declared cured after treatment).
4. Pregnant or breastfeeding women.
5. Positive test for anti-HIV antibodies.
6. Active HBV or HCV infection considered clinically inappropriate for study participation by the investigator.
7. Uncontrolled central nervous system (CNS) metastases (note: patients with treated and stable brain metastases for ≥30 days prior to screening are eligible).
8. Any surgery, radiotherapy, or systemic anticancer therapy within 3 weeks prior to CT-SP administration.
9. Participation in another interventional clinical trial and receipt of any investigational drug within 3 weeks prior to CT-SP administration.
10. Known hypersensitivity or contraindication to: Cyclophosphamide, Fludarabine, Interleukin-2 (IL-2), CT-SP excipients: 5% human serum albumin, sterile saline, 5% DMSO
11. Unresolved toxicity from prior therapy not recovered to Grade ≤1 (per NCI CTCAE v5.0), except for clinically non-significant events such as alopecia.
12. Receipt of systemic immunosuppressive therapy (including corticosteroids) within 10 days prior to tumor tissue collection for CT-SP manufacturing (exceptions: local/inhaled steroids; systemic corticosteroids ≤ prednisolone 20 mg/day equivalent may be permitted at investigator discretion).
13. Clinically significant cardiovascular disease, including but not limited to:

    Uncontrolled hypertension (systolic BP > 180 mmHg and/or diastolic BP > 100 mmHg), Unstable angina, Pulmonary embolism, Cerebrovascular accident, Valvular heart disease, Congestive heart failure (NYHA Class III or IV), Myocardial infarction or significant arrhythmia within 24 weeks prior to screening
14. Known contraindications to dopamine or other pressor agents.
15. Other serious comorbid medical conditions that may interfere with study participation, as determined by the investigator.
16. Active or severe infection requiring hospitalization or intravenous antibiotics, deemed unsuitable for participation by the investigator.
17. Significant psychiatric illness that, in the investigator's opinion, may affect subject compliance or study conduct.
18. Subjects with autoimmune or inflammatory disorders, where the investigator deems abnormal autoantibody test results to be clinically relevant.
19. Any other condition not listed above that the investigator considers to make the subject ineligible for participation.
20. Subjects determined to be unsuitable for participation based on the anticipated manufacturing timeline and logistics of CT-SP.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-05-28 (Estimated); Study Completion 2029-05-28 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation | up to 6 months after TIL administration
  Incidence of tumor infiltration lymphocyte (CT-SP) treatment Adverse Events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Overall Response Rate | Up to 60months
  modified Recist v1.1
Duration of Response | Up to 60months
  modified Recist v1.1
Disease Control Rate | Up to 60months
  modified Recist v1.1
Progression Free Survival | Up to 60months
  modified Recist v1.1
Overall Survival | Up to 60months
  modified Recist v1.1

IPD SHARING:
Plan to Share IPD: No